CLINICAL TRIAL: NCT04319315
Title: Impact of Social Media on Knowledge Dissemination Between Physicians During COVID-19 Virus Outbreak
Brief Title: Social Media Effect on Knowledge Dissemination During COVID-19 Virus Outbreak
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: AssiutU-3-2020
Record Dates: First submitted 2020-03-16; First posted 2020-03-24 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: COVID-19
Keywords: Corona Virus; Social Media; Physician; Knowledge
MeSH Terms: conditions — COVID-19 | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey — online survey

SUMMARY:
The recent COVID-19 outbreak is very challenging as data are distributed instantly on the data are very rapidly distributed through professional and non professional sources which may impact the management of the disease

DETAILED DESCRIPTION:
The investigators are conducting a survey between the physicians to study the effect and practice of received knowledge disseminated through social media .

the survey will be distributed through internet and data will be collected and analyzed

ELIGIBILITY:
Inclusion Criteria:

* Medical Physicians in Middle East area

Exclusion Criteria:

* none

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: the study survey will be distributed through email to medical physicians in our territory
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-03-11 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-16 (Estimated)

PRIMARY OUTCOMES:
Number of physicians affected by social media measured by online survey designed to measure the influence of social media on medical practice | one month
  the survey will be send and received online and data will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Aliae Mohamed-Hussein, Principal Investigator — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No